CLINICAL TRIAL: NCT04490785
Title: Characterization of Postoperative Myocardial Lesions by Cardiac MRI and Anatomo-biological Correlations With Serum Troponin in Cardiac Surgery.
Brief Title: Mri characterIzation of Troponin Elevation After Cardiac Surgery
Acronym: MITEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0020
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Cardiac surgery; Cardiopulmonary bypass; ischemia reperfusion; Cardiac magnetic resonance imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients under aortic surgery with CPB (Experimental): Patients under aortic surgery with CPB will have MRI and postoperative dosage of released troponin
  Interventions: Procedure: MRI; Biological: Postoperative dosage of released troponin

INTERVENTIONS:
Procedure: MRI — 1 MRI 5 days after surgery (-1; +4 days), with intravenous administration of gadolinium
Biological: Postoperative dosage of released troponin — Dosage of troponin I Hs H4, H8, H12, H24, H48, and H72 after the aortic cross-unclamping.

SUMMARY:
Cardiac surgery under cardiopulmonary bypass (CPB) induces myocardial ischemia-reperfusion injury. This myocardial attack is a well-identified independent prognostic factor of postoperative morbidity and mortality. The quantification of these myocardial lesions by the postoperative plasma release of troponin has proven its diagnostic and prognostic value.

Cardiac magnetic resonance imaging (MRI) can accurately measure and characterize the size of myocardial lesions. These lesions are associated with a poor prognosis. MRI can also characterize myocardial edema secondary to ischemia-reperfusion which has not yet been studied in the context of CPB. It is therefore necessary, in a mechanistic approach, to quantify the respective share of necrosis, edema and reperfusion lesions during cardiac surgery under CPB in order to better understand these phenomena and to propose effective strategies for the prevention of these myocardial lesions.the relationship between the postoperative release of troponin and the amount of myocardial necrosis and edema measured by cardiac MRI will be assessed.The hypothesis is to demonstrate a positive correlation between imaging and biology in order to better understand the perioperative myocardial lesion processes.

This is an interventional study prospective, exploratory, in cardiac imaging, non-comparative and single-center, including 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Aortic valve surgery with CEC: aortic valve replacement, Bentall, Tirone-David, Wheat with foreseeable clamping time of at least 40 minutes.
* Informed consent signed

Exclusion Criteria:

* Emergency surgery
* Other unconventional heart surgery
* Aorto-coronary bypass associated with surgery
* History of myocardial infarction or severe coronary artery disease, non-valvular hypertrophic cardiomyopathy (MHC) (primary MHC type, Amyloidosis) and myocarditis
* Preoperative alteration of systolic function of the left ventricle (LVEF <40%)
* Presence of a contraindication to cardiac MRI (claustrophobia, pacemaker or cardiac defibrillator, metallic body, hypersensitivity to gadolinium)
* Patients with a glomerular filtration rate (GFR) <30 ml / min
* Patients with permanent atrial fibrillation (ACFA) cardiac arrhythmia
* Patients treated with anthracyclines
* Pregnant and / or lactating woman
* Patient under legal protection
* Patient not benefiting from a social security system
* Patient participating in another clinical study that may interfere with the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
correlation between cardiac MRI and the AUC of postoperative plasma released hsTnI. | 5 days
  Correlation between the AUC of plasma hsTnI levels measured during the first 72 hours postoperatively (sequential basal assays then 4, 8, 12, 24, 48 and 72 hours after aortic unclamping) and the mass in grams of myocardial necrosis measured by the late enhancement in cardiac MRI on D5 postoperative. Correlations between MRI anatomical data and biological or ultrasound data will be assessed with the Pearson or Spearman correlation coefficient according to the distribution of variables and linear regression.

SECONDARY OUTCOMES:
Relationship between peak serum hsTnI and mass in grams of necrosis on MRI. | 5 days
  Correlation between highest serum value recorded for each patient within 72 hours and the mass in grams of myocardial necrosis measured by the late enhancement in cardiac MRI on D5 postoperative.
AUC / serum peak hsTnI relationship and relative size of the necrosis on MRI | 5 days
  Correlation between the AUC of plasma hsTnI levels measured during the first 72 hours postoperatively (sequential basal assays then 4, 8, 12, 24, 48 and 72 hours after aortic unclamping) and percentage of left ventricular mass. Correlation between highest serum value recorded for each patient within 72 hours and percentage of left ventricular mass.
Relationship of hsTnI levels at 24 hours after aortic unclamping and the mass in grams of necrosis on MRI. | 5 days
  Correlation between the AUC of plasma hsTnI levels measured at 24 hours after aortic unclamping and the mass in grams of myocardial necrosis measured by the late enhancement in cardiac MRI on D5 postoperative.
AUC / peak serum hsTnI relationship and intensity of edema | 5 days
  Correlation between the AUC of plasma hsTnI levels measured during the first 72 hours postoperatively (sequential basal assays then 4, 8, 12, 24, 48 and 72 hours after aortic unclamping) and intensity of edema at MRI. Correlation between highest serum value recorded for each patient within 72 hours and intensity of edema at MRI
AUC / hsTnI serum peak relationship and the presence of microvascular obstruction lesions on MRI on postoperative D5 | 5 days
  Correlation between the AUC of plasma hsTnI levels measured during the first 72 hours postoperatively (sequential basal assays then 4, 8, 12, 24, 48 and 72 hours after aortic unclamping) and the presence of microvascular obstruction lesions on MRI on postoperative D5.
  Correlation between highest serum value recorded for each patient within 72 hours and the presence of microvascular obstruction lesions on MRI on postoperative D5.
Relation of functional and anatomical parameters evaluated by cardiac MRI on postoperative D5. | 5 days
  Tele-diastolic volume / ventricular mass, LVEF on MRI on postoperative D5.
Correlations between clamping time and CEC and the size of the reperfusion lesions visible on MRI on D5 postoperative | 5 days
  Correlation between clamping time and the size of the reperfusion lesions visible on MRI on D5 postoperative.
  Correlation between CEC time and the size of the reperfusion lesions visible on MRI on D5 postoperative.
Exploratory evaluation of the kinetic profile of AUC with the type of lesion found on cardiac MRI (early peak, versus late peak). | 5 days
  Correlation between the kinetic profile of AUC and the type of lesion found on MRI on D5 postoperative.
Relation of functional and anatomical parameters of the right ventricle in 4 cavities and small axis (tele-diastolic volume, FEVD) evaluated by cardiac MRI on D5 postoperative. | 5 days
  Correlation between the right ventricle in 4 cavities and small axis (2 differents measures) on MRI on D5 postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fellahi JL, Ferraris A, Chiari P, Varillon Y, De Bourguignon C, Mewton N. High-Sensitivity Troponin I Release After Aortic Surgery: A Mechanistic Approach with Contrast-Enhanced Magnetic Resonance Imaging (the MITEC Study). Anesth Analg. 2025 Jan 1;140(1):228-230. doi: 10.1213/ANE.0000000000007165. Epub 2024 Oct 15. No abstract available. PMID 39466631